CLINICAL TRIAL: NCT01004640
Title: Molecular and Cytogenetic Monitoring of CML - A Mandatory Companion to CALGB 19804
Brief Title: Study of Blood and Bone Marrow Samples in Patients With Chronic Myelogenous Leukemia Enrolled on a CALGB Clinical Trial
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-29801; U10CA031946 (NIH); U10CA180821 (NIH); CDR0000078595 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Leukemia
Keywords: chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Blotting, Southern; Cytogenetic Analysis; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Peripheral blood samples and bone marrow aspirates are collected at baseline and at 3, 6, and 9 months after starting therapy. If patient continues to receive protocol treatment after 9 months, additional peripheral blood samples are collected every 6 months and bone marrow aspirates are taken annually. In the event of disease progression (blast crisis), an additional peripheral blood sample and bone marrow aspirate are collected.
  Samples are examined by quantitative Southern blot analysis with probes to BCR, quantitative reverse transcriptase-polymerase chain reaction analysis for BCR/ABL fusion transcripts, and cytogenetic analysis.
  Interventions: Genetic: DNA analysis; Genetic: Southern blotting; Genetic: cytogenetic analysis; Genetic: polymerase chain reaction

INTERVENTIONS:
Genetic: DNA analysis
Genetic: Southern blotting
Genetic: cytogenetic analysis — Correlative studies
  Other Names: Laboratory Biomarker Analysis
Genetic: polymerase chain reaction

SUMMARY:
RATIONALE: Studying samples of blood and bone marrow from patients with cancer may help doctors identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood and bone marrow samples in patients with chronic myelogenous leukemia enrolled on a CALGB clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* Monitor molecular response rates of patients receiving treatment for chronic myelogenous leukemia by quantitative reverse transcription polymerase chain reaction (RT-PCR) and quantitative Southern blot monitoring of blood samples.
* Compare quantitative RT-PCR and quantitative Southern blot results with marrow cytogenetics at the time of complete molecular response in these patients.
* Monitor the frequency of residual disease in patients who achieve a complete blood Southern blot and marrow cytogenetic response (eradication of BCR/ABL by Southern blot and absence of the Philadelphia chromosome by cytogenetics).

OUTLINE: Peripheral blood samples and bone marrow aspirates are collected at baseline and at 3, 6, and 9 months after starting therapy. If patient continues to receive protocol treatment after 9 months, additional peripheral blood samples are collected every 6 months and bone marrow aspirates are taken annually. In the event of disease progression (blast crisis), an additional peripheral blood sample and bone marrow aspirate are collected.

Samples are examined by quantitative Southern blot analysis with probes to BCR, quantitative reverse transcriptase-polymerase chain reaction analysis for BCR/ABL fusion transcripts, and cytogenetic analysis.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic myelogenous leukemia (CML)
* Concurrent enrollment on a CALGB treatment protocol for newly diagnosed or previously treated CML (e.g, CLB-19804)

  * Must not have initiated study therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PATIENTS ENTERED ONTO CALGB TREATMENT STUDIES FOR CML
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 1998-12-15 (Actual); Primary Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Distribution response | Up to 1.5 years
Distribution of cytogenetic response | Up to 1.5 years
Distribution of RT-PCR response or Southern blot response | Up to 1.5 years
Frequency of residual disease in patients who have achieved a complete response | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, MD, Study Chair — University of Chicago
Locations (161):
- United States (161):
  - Naval Medical Center - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health Services, Newark, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Saint Francis Hospital - Wilmington, Wilmington, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Assocation, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois Oncology Limited, Granite City, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Hopedale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Illinois CancerCare- Ottawa Clinic, Ottawa, Illinois
  - Ottwa Regional Hospital and Healthcare, Ottawa, Illinois
  - Illinois CancerCare- Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare- Peoria, Peoria, Illinois
  - Illinois Oncology Research Association-CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare- Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare- Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Sarah Culberston Memorial Hospital, Rushville, Illinois
  - Illinois CancerCare- Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Saint Joseph Regional Medical Center - Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consrtium, South Bend, Indiana
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Eastern Maine Medical Center, Bangor, Bangor, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Commonwealth Hematology Oncology PC-Worcester, Worcester, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Missouri Cancer Associates, Columbia, Missouri
  - Veterans Administration, Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - University of Missouri - Ellis Fischel,, Columbia, Missouri
  - Capital Regional Medical Center, Jefferson City, Missouri
  - Lakeland Hospital, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Valley Regional, Claremont, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Weeks Memorial Hospital, Lancaster, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Alice Peck Day Memorial Hospital, Lebanon, New Hampshire
  - Frisbie Hospital, Rochester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Queens Hospital Center, Jamaica, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Oswego Hospital, Oswego, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, Syracuse, New York
  - Saint Joseph's Hospital Health Center, Syracuse, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Mission Hospital-Saint Joseph Campus, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Lenoir Memorial Hospital, Kinston, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Cancer Centers of the Carolinas-Green Medial Oncology, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Central Vermont Medical Center/ National Life Cancer Treatment, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - North Country Health, Newport, Vermont
  - Northeastern, Saint Johnsbury, Vermont
  - Springfield Hospital, Springfield, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - Danville Regional Medical Center, Danville, Virginia